CLINICAL TRIAL: NCT04403594
Title: Functional Intermuscular Reduction of SpasTicity in MS (MS-FIRST)
Brief Title: Functional Intermuscular Reduction of Spasticity
Acronym: MS-FIRST
Status: Completed | Type: Observational
Sponsor: University of Oklahoma (Other)
Collaborators: Oklahoma Medical Research Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 19-21
Record Dates: First submitted 2020-05-13; First posted 2020-05-27 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Dry Needling

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MS with spasticity of one lower extremity: A person diagnosed with Multiple Sclerosis and spasticty of one lower extremity. The person must be able to walk 25 feet and cannot have had Botox in the lower extremity on the last 6 months.
  Interventions: Other: dry needling

INTERVENTIONS:
Other: dry needling — dry needling followed by functional electrical stimulation and treadmill training
  Other Names: functional electrical stimulation

SUMMARY:
Investigators will use muscular dry needling in the calf of one lower extremity, followed by treadmill training with functional electrical stimulation.

DETAILED DESCRIPTION:
This study will be the first to combine a novel two-pronged approach to the management of spasticity (tightness of the muscle) in the calf muscles. First, investigators will decrease spasticity in an innovative way through dry needling. Second, investigators will follow this spasticity reduction technique using external electrical stimulation applied to the calf, while the participant walks on a harnessed treadmill (for safety). The investigators believe modulating tone in the calf with dry needling will allow for improved strength with electrical stimulation, while simultaneously improving the efficiency of the muscles during walking. The investigators hypothesize that decreasing spasticity will result in enhanced gait efficiency, and lower fatigue, all while allowing the participant to meet their personal mobility goals.10 The investigators are proposing an innovative study design. Assessing changes in muscle spasticity using electromyography and the Modified Ashworth scale before and after each portion of our two-pronged intervention will enable them to understand the immediate effects of dry needling, as well as the combined effects of function electrical stimulation with with treadmill training. Following the intervention assessments with pre-post functional tests will allow us to determine long term changes. This proposal offers a unique approach to management of spasticity in people with Multiple Sclerosis (MS), with the advantage of being minimally invasive and inexpensive. Results of this pilot study will inform the potential use in MS, and will allow for a larger study examining optimal intervention parameters for future use.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of MS based on MRI
2. Ability walk 25 feet
3. Spasticity of one lower extremity

Exclusion Criteria:

1. Blood clot within the last 6 months
2. Bleeding disorder
3. Active cancer
4. Botox in the lower extremities within 6 months

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: People with a diagnosis of MS and spasticity
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2019-08-19 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-18 (Actual)

PRIMARY OUTCOMES:
6 minute walk test | up to 7 weeks
  distance walked over 6 minutes assessed at the start of the study and after 6 weeks.
25-foot walk | up to 7 weeks
  time to walk 25 feet assessed at the start of the study and after 6 weeks.
Berg Balance Scale | up to 7 weeks
  Balance test conducted at the start of the study and after 6 weeks.
Modified Fatigue Impact Scale | up to 7 weeks
  patient-reported questionnaire collected at the start of the study and after 6 weeks.
Toe taps on force plate | up to 7 weeks
  number of toe taps in 10 seconds counted at the start of the study and after 6 weeks.
EMG data of both lower extremities | up to 7 weeks
  Electromyography (EMG) will be conducted at the start of the study and after 6 weeks. EMG is an electrodiagnostic technique for evaluating and recording the electrical activity produced by skeletal muscles. This is completed using electrodes that are placed on the skin, which detects the electric potential generated by muscle cells when these cells are electrically or neurologically activated. These action potentials are measured and recorded on a computer.

CONTACTS AND LOCATIONS:
Overall Officials: Shirley James, PhD, Principal Investigator — University of Oklahoma
Locations (1):
- Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No